CLINICAL TRIAL: NCT04831632
Title: Diagnostic Performance Assessment of Qualitative Ifobt and Various Quantitative Ifobt Cut-off Points for Advanced Neoplastic Wound Screening in an Argentine Patient Cohort
Brief Title: Diagnostic Performance Assessment of Qualitative Ifobt and Quantitative Ifobt for Advanced Neoplastic
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: CECILIA CURVALE (Other)
Collaborators: Ministry of Public Health, Argentina (Other Government)
Responsible Party: Sponsor-Investigator, CECILIA CURVALE, Clinical Investigator, Hospital El Cruce
Organization: Hospital El Cruce (Other)
Other Study IDs: 091/2020
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Colorectal Neoplasms
Keywords: screening; colorectal cancer; fecal immunochemical test; FIT accuracy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- people aged 50-75: men and women aged 50-75 who belong to Hospital El Cruce's coverage area and do not have personal history of colorectal cancer or inflammatory bowel disease, personal or family history of syndromes of predisposition to known cancers, or family history of colorectal cancer in a first-degree relative aged less than 60
  Interventions: Diagnostic Test: quantitative and qualitative iFOBTs

INTERVENTIONS:
Diagnostic Test: quantitative and qualitative iFOBTs — They will have their qualitative and quantitative iFOBTs done within the week prior to the VCC study completion. The reading of both of them will be done in Hospital El Cruce's laboratory. The result of the qualitative iFOBT will have two valid expressions: positive or negative.The result of the quantitative iFOBT will be expressed as µg from hemoglobin per gram of fecal matter through the use of automatized equipment for laboratory analysis.

SUMMARY:
In Argentina, there is vast experience in qualitative iFOBT population screening that is part of the CRC Prevention and Early Detection National Program. The screening's cut-off point is at 50 ng/mL buffer. Its positivity rate for 2019 has been an average of 26.15%, over the double of the one reported in the international literature (7.5-11%) for this cut-off point (1). There are no studies that assess such technology and suggest an appropriate cut-off point for this population. The goal of this study is to assess the diagnostic performance of the qualitative iFOBT used in the present and the quantitative iFOBT with various cut-off points for advanced neoplastic wound screening (colorectal cancer and advanced adenoma) in an Argentine patient cohort.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 50-75
* Hospital El Cruce's coverage area and

Exclusion Criteria:

* those that have taken part in a previous VCC screening in the 5 past years or in a CRC screening program the year before the recruitment
* personal history of colorectal cancer or inflammatory bowel disease, personal or family history of syndromes of predisposition to known cancers, or family history of colorectal cancer in a first-degree relative aged less than 60
* those refuse to sign the consent form to take part in this study

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: people who belong to Hospital El Cruce's coverage area
Sampling Method: Probability Sample
Enrollment: 630 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
diagnostic performance | 2 years
  To determine the diagnostic performance of the quantitative iFOBT with various cut-off points and the qualitative iFOBT, compared to the VCC, when detecting advanced colon neoplasms.

SECONDARY OUTCOMES:
qualitative iFOBT positivity rate | 2 years
  To set the qualitative iFOBT positivity rate at 50 ng/mL in a controlled Argentine cohort.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital El Cruce, San Juan Bautista, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided